CLINICAL TRIAL: NCT06857227
Title: A Randomized Controlled Phase l Clinical Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics/Pharmacodynamics of GNC-038 Tetra-specific Antibody Injection in Rheumatoid Arthritis
Brief Title: A Study of GNC-038 Tetra-specific Antibody Injection in Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GNC-038-107
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNC-038 (Experimental): Participants receive GNC-038 in the first cycle. Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-038
- Placebo (Placebo Comparator): The control group will be set up in phase Ib, participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GNC-038 — Administration by intravenous infusion. Once a week (IV, QW), twice in total.
  Arms: GNC-038
Drug: Placebo — The control group will be set up in phase Ib, and an appropriate dose will be selected based on phase Ia data.
  Arms: Placebo

SUMMARY:
This study is a randomized controlled phase I clinical study with safety, efficacy, and pharmacokinetic/pharmacodynamic characteristics in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
This study is divided into a phase Ia study and a phase Ib study. The phase Ib study has a randomized controlled design with a placebo control group. The phase Ia study has a single-arm design, and the phase Ib study will be carried out on the basis of the Phase Ia study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can understand the informed consent form, voluntarily participate in and sign the informed consent form;
2. No gender limit;
3. Age: ≥18 years old and ≤75 years old;
4. Life expectancy greater than 6 months;
5. Patients diagnosed with rheumatoid arthritis according to 1987 or 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria;
6. Patients were moderately to severely active RA at the time of screening;
7. A stable standard-of-care regimen was maintained for at least 30 days before the first dose;
8. Previous treatment with antirheumatic drugs other than MTX: Leflunomide should be discontinued at least 8 weeks before the start of study treatment or cholestyramine should be used for 14 days;
9. Erythrocyte sedimentation rate (ESR) > 28mm/hr or C-reactive protein (CRP) > 10mg/L;
10. Positive rheumatoid factor and/or anti-cyclic citrullinated peptide antibodies;
11. There were CD19+ B cells in the peripheral blood of the patient;
12. Diagnosis of rheumatoid arthritis (RA) more than 6 months;
13. The organ function level before the first administration met the requirements;
14. Fertile female subjects or male subjects with fertile partners must use highly effective contraception from 7 days before the first dose until 24 weeks after the termination of treatment and should commit not to donate eggs (eggs, oocytes)/sperm for assisted reproduction for 1 year after the last study treatment. Female subjects of childbearing potential must have a negative serum/urine pregnancy test within 7 days before the first dose;
15. Participants were able and willing to comply with protocol-specified visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Confirmed diagnosis of another autoimmune rheumatic disease;
2. B cell-targeted therapy agents administered within 6 months before GNC-038 treatment;
3. Received CAR-T therapy within 6 months before GNC-038 treatment;
4. Use of anti-TNF drugs within 8 weeks before administration;
5. Use of any JAK inhibitor within 2 weeks before dosing;
6. Antimalarial drugs, sulfasalazine, penicillamine, etc. were used within 4 weeks before the drug administration;
7. Use of phytochemicals within 4 weeks before administration;
8. The use of other biological agents or other non-B cell depleting clinical investigational drugs before drug administration did not exceed 5 half-lives;
9. Received an intra-articular injection within 4 weeks before study entry;
10. Receipt of any investigational drug within 28 days before dose or within 5 half-lives of the investigational drug;
11. ACR functional class IV or bedridden/wheelchair-bound;
12. History of major organ transplantation or hematopoietic stem cell/bone marrow transplantation;
13. Presence of: 1) active hepatitis B at screening; 2) hepatitis C or HIV infection; 3) syphilis infection;
14. A history of any cardiovascular disease described in the protocol within 6 months before screening;
15. Poorly controlled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg);
16. Prolonged QT interval at rest (QTcf > 450 msec in men or > 470 msec in women);
17. A history of ≥ grade 2 bleeding within 30 days before screening or the need for long-term continuous anticoagulant therapy;
18. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of GNC-038;
19. Women who are pregnant or breastfeeding;
20. Having a history or evidence of suicidal thoughts within 6 months before signing ICF, which is considered by the researcher to be a significant risk of suicide;
21. Diagnosed with malignant tumor within 5 years before signing ICF;
22. Other situations of poor compliance, unwillingness or inability to comply with the study protocol as judged by the investigator;
23. History of splenectomy;
24. Investigators considered a history of alcohol or drug abuse in the 12 months before screening;
25. Any active infection requiring systemic antibiotic treatment within 2 weeks before or during screening;
26. A history of severe and/or disseminated viral infection;
27. Active M. tuberculosis infection may be present.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to approximately 28 days
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) or Maximum administered dose (MAD) | Up to approximately 28 days
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle.
Phase Ia: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-038. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-038.
Phase Ia: Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of GNC-038 will be investigated.
Phase Ia: Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of GNC-038 will be investigated.
Phase Ia: T1/2 | Up to approximately 24 months
  Half-life (T1/2) of GNC-038 will be investigated.
Phase Ia: AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
Phase Ia: CL (Clearance) | Up to approximately 24 months
  CL in the serum of GNC-038 per unit of time will be investigated.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-038.
Phase Ib: Proportion of patients meeting ACR20 remission criteria | Up to approximately 24 months
  Proportion of patients meeting ACR20 remission criteria will be investigated.

SECONDARY OUTCOMES:
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-GNC-038 antibody (ADA) will be investigated.
Phase Ia: Receptor Occupancy (RO) | Up to approximately 24 months
  Receptor Occupancy (RO) will be investigated.
Phase Ib: Change from baseline in quality of life (SF-36) | Up to approximately 24 months
  Change from baseline in quality of life (SF-36) will be investigated.
Phase Ib: Change from baseline in DAS28 CRP | Up to approximately 24 months
  Change from baseline in DAS28 CRP will be investigated.
Phase Ib: Proportion of patients meeting ACR50 response criteria | Up to approximately 24 months
  Proportion of patients meeting ACR50 response criteria will be investigated.
Phase Ib: Proportion of patients meeting ACR70 response criteria | Up to approximately 24 months
  Proportion of patients meeting ACR70 response criteria will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China